CLINICAL TRIAL: NCT04556825
Title: Prospective Randomized Controlled Study on Arthroscopic Treatment Combined With PRP Injection for Refractory Elbow Epicondylitis
Brief Title: Arthroscopic Treatment Combined With PRP Injection for Refractory Elbow Epicondylitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Yi Lu, Director of Sports Medicine Service of Beijing Jishuitan hospital, Beijing Jishuitan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YiL
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: PRP; Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Arthroscopic treatment with PRP injection
  Interventions: Drug: PRP
- Control group (Placebo Comparator): Arthroscopic treatment with normal saline injection
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: PRP — After the arthroscopic operation was completed, a local PRP with 4ml was injected
  Arms: Study group
Drug: normal saline — After the arthroscopic operation was completed, a local normal saline injection with same ml was performed
  Arms: Control group

SUMMARY:
This study is a prospective randomized controlled study of different arthroscopic treatments for refractory external humeral epicondylitis combined with platelet rich plasma (PRP) injection. The patients with intractable external humeral epicondylitis were randomly divided into groups before the operation. After the arthroscopic operation was completed, they were divided into a local PRP injection group and a control group (normal saline) to perform additional operations on the damaged tendons, each for up to half a year after the operation. In different time periods, the quantitative and qualitative indicators including pain, functional score, muscle strength, MRI performance, etc. were compared between groups at the same time period to evaluate the difference in the effect of arthroscopic treatment combined with PRP on the treatment of damaged tendons. Determine the effectiveness of PRP. At the same time, in the process of arthroscopic treatment, look for risk factors that affect the curative effect of intractable external humeral epicondylitis, as well as the causes and prevention of common complications.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed patients with refractory external humeral epicondylitis (preoperative MRI confirmed loss of ECRB integrity) patients who have received non-surgical treatment with poor efficacy
* Young and middle-aged patients aged 20 to 60, who have not previously received local injection therapy
* Voluntarily accept randomized controlled grouping, cooperate with treatment and follow up patients
* No other comorbidities or medical diseases affect the surgical patients
* Unilateral disease

Exclusion Criteria:

* Early patients who have not received standard non-surgical treatment
* Patients who have received hormone injections or "small needle knife therapy" and other invasive procedures within three months before surgery, poor skin conditions, and local infections
* Elderly people older than 60 years old and patients younger than 20 years old
* Unable to accept randomization, insufficient follow-up time or lost to follow-up
* Bilateral disease
* Combined immune disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Mayo Elbow Performance Score | 3, 6 weeks and 3, 6, 12, 24 months postoperatively
  A score used to evaluated the elbow function, higher scores mean a better outcome.

SECONDARY OUTCOMES:
Integrity of the tendon in MRI | 3, 6, 12, 24 months postoperatively
  MRI was performed to identify the status of the tendon
Disability of the Arm, Shoulder, and Hand (DASH) | 3, 6 weeks and 3, 6, 12, 24months postoperatively
  A score used to evaluated the elbow function, higher scores mean a worse outcome.
Patient-Rated Tennis Elbow Evaluation (PRTEE) scale | 3, 6 weeks and 3, 6, 12, 24months postoperatively
  A score used to evaluated the elbow function, higher scores mean a worse outcome
scoring system of Verhaar | 3, 6 weeks and 3, 6, 12, 24months postoperatively
  A score used to evaluated the elbow function, higher scores mean a better outcome
visual analog scale (VAS) | 3, 6 weeks and 3, 6, 12, 24months postoperatively
  A score used to evaluated the elbow function, higher scores mean a better

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lu, Principal Investigator — Sports Medicine Service, Beijing Jishuitan hospital
Locations (1):
- Beijing Jishuitan hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li S, Yang G, Chen R, Li X, Lu Y. Use of Adjunctive Platelet-Rich Plasma for Healing During Arthroscopic Release and Repair for Recalcitrant Lateral Epicondylitis: A Prospective, Double-Blind, Randomized Controlled Trial. Am J Sports Med. 2025 Jul;53(8):1817-1825. doi: 10.1177/03635465251341458. Epub 2025 May 31. PMID 40448507